CLINICAL TRIAL: NCT06602089
Title: Superiority of Finger-sensor Over Oscillometric Arterial Pressure Monitoring in Patients Having Non-cardiac Surgery: the Prospective Observational PERCEPTION Study
Brief Title: Superiority of Finger-sensor Monitoring: a Prospective Observational Study
Acronym: PERCEPTION
Status: Completed | Type: Observational
Sponsor: University of Hamburg-Eppendorf (Other)
Responsible Party: Principal Investigator, Dr. Alina Bergholz, Principal Investigator, University of Hamburg-Eppendorf
Other Study IDs: 2024-101274-BO-ff
Record Dates: First submitted 2024-09-08; First posted 2024-09-19 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Blood Pressure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: Arterial pressure monitoring — We will record intraarterial arterial pressure, finger-sensor arterial pressure and oscillometric arterial pressure in all included patients.

SUMMARY:
This is an observational study investigating whether finger-sensor arterial pressure monitoring is superior to oscillometric arterial pressure monitoring in patients having non-cardiac surgery. Specifically, the investigators will test the hypothesis that the agreement between finger-sensor arterial pressure measurements and intraarterial arterial pressure measurements (mean arterial pressure, systolic arterial pressure, and diastolic arterial pressure) is better than the agreement between oscillometric mean arterial pressure measurements and intraarterial mean arterial pressure measurements in patients having low- to moderate-risk non-cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years
* scheduled for elective low- to moderate-risk non-cardiac surgery with general anesthesia
* planned intraarterial arterial pressure monitoring

Exclusion Criteria:

* systolic arterial pressure interarm differences >20 mmHg
* heart rhythms other than sinus rhythm
* contraindications for finger-sensor arterial pressure monitoring (e.g., arteriovenous shunts, Raynaud's disease)
* pregnant patients.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients ≥18 years scheduled for elective low- to moderate-risk non-cardiac surgery with general anesthesia in whom intraarterial arterial pressure monitoring is planned
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2024-09-09 (Actual); Primary Completion 2025-06-26 (Actual); Study Completion 2025-06-26 (Actual)

PRIMARY OUTCOMES:
Difference in the agreement between finger-sensor arterial pressure measurements and intraarterial arterial pressure measurements, and the agreement between oscillometric arterial pressure measurements and intraarterial arterial pressure measurements | During surgery
  To investigate whether the agreement between finger-sensor arterial pressure measurements and intraarterial arterial pressure measurements (mean arterial pressure, systolic arterial pressure, and diastolic arterial pressure) is better than the agreement between oscillometric arterial pressure measurements and intraarterial arterial pressure measurements, we will perform Bland-Altman analyses.

SECONDARY OUTCOMES:
Classification of measurement differences between finger-sensor arterial pressure measurements and intraarterial arterial pressure measurements according to their clinical importance | During surgery
  To classify measurement differences (mean arterial pressure and systolic arterial pressure) between finger-sensor arterial pressure measurements and intraarterial arterial pressure measurements according to their clinical importance, we will perform error grid analyses.
Classification of measurement differences between oscillometric arterial pressure measurements and intraarterial arterial pressure measurements according to their clinical importance | During surgery
  To classify measurement differences (mean arterial pressure and systolic arterial pressure) between oscillometric arterial pressure measurements and intraarterial arterial pressure measurements according to their clinical importance, we will perform error grid analyses.
Ability of finger-sensor arterial pressure monitoring to track arterial pressure changes compared to intraarterial arterial pressure monitoring | During surgery
  To investigate the ability of finger-sensor arterial pressure monitoring to track arterial pressure changes (mean arterial pressure, systolic arterial pressure, and diastolic arterial pressure) compared to intraarterial arterial pressure monitoring, we will compute four-quadrant plots and calculate the concordance rate.
Ability of oscillometric arterial pressure monitoring to track arterial pressure changes compared to intraarterial arterial pressure monitoring | During surgery
  To investigate the ability of oscillometric arterial pressure monitoring to track arterial pressure changes (mean arterial pressure, systolic arterial pressure, and diastolic arterial pressure) compared to intraarterial arterial pressure monitoring, we will computer four-quadrant plots and calculate the concordance rate.

CONTACTS AND LOCATIONS:
Overall Officials: Alina Bergholz, MD, Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (1):
- Department of Anesthesiology, Center of Anesthesiology and Intensive Care Medicine, University Medical Center Hamburg-Eppendorf, Hamburg, Germany